CLINICAL TRIAL: NCT05109390
Title: A Three-Part Phase 1 Study to Evaluate the Potential Drug Interaction Between ACH-0144471 and Cyclosporine, Tacrolimus, Antacids, and Omeprazole in Healthy Adult Subjects
Brief Title: A Study of the Drug Interactions Between Danicopan and Cyclosporine, Tacrolimus, Antacids, and Omeprazole in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Achillion, a wholly owned subsidiary of Alexion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ACH471-014
Record Dates: First submitted 2021-09-09; First posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Healthy
Keywords: Danicopan; ALXN2040; ACH-0144471; Drug Interaction; Cyclosporine; Tacrolimus; Antacids; Omeprazole
MeSH Terms: interventions — danicopan; rhoA GTP-Binding Protein; Cyclosporine; Tacrolimus; Calcium Carbonate; Antacids; aluminum hydroxide, magnesium hydroxide, simethicone drug combination; Gelusil; Omeprazole

STUDY DESIGN:
Intervention Model Description: This was a 3-part study, each part is a fixed-sequence with 2 periods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Danicopan plus Cyclosporine (Experimental): Participants (N=14) received danicopan and cyclosporine in a fixed sequence over 2 periods:
  Treatment A (Period 1): 300 milligrams (mg) cyclosporine administered on Day 1.
  Treatment B (Period 2): 200 mg danicopan administered 3 times daily (TID) on Days 1-7 with 300 mg cyclosporine coadministered on Day 5.
  There was a washout period of 3 days between the dose of cyclosporine in Period 1 and the first dose of danicopan in Period 2.
  Interventions: Drug: Danicopan; Drug: Cyclosporine
- Part 2: Danicopan plus Tacrolimus (Experimental): Participants (N=28) received danicopan and tacrolimus in a fixed sequence over 2 periods:
  Treatment C (Period 1): 2 mg tacrolimus administered on Day 1.
  Treatment D (Period 2): 200 mg danicopan administered TID on Days 1-10 with 2 mg tacrolimus coadministered on Day 5.
  There was a washout period of 7 days between the dose of tacrolimus in Period 1 and the first dose of danicopan in Period 2.
  Interventions: Drug: Danicopan; Drug: Tacrolimus
- Part 3: Danicopan plus Antacids and Omeprazole (Experimental): Participants (N=30) received danicopan, calcium carbonate, aluminum/magnesium hydroxide/simethicone, and omeprazole in fixed sequences over 2 periods:
  Treatment E1 (Period 1): 200 mg danicopan administered TID on Days 1-4. Treatment E2 (Period 1): 200 mg danicopan coadministered with 1 gram calcium carbonate on Day 5.
  Treatment F1 (Period 1): 200 mg danicopan administered TID on Days 1-4. Treatment F2 (Period 1): 200 mg danicopan coadministered with 200 mg aluminum hydroxide/200 magnesium hydroxide/25 mg simethicone on Day 5.
  Note: Participants were randomized in a 1:1 ratio to receive either Treatment E2 or F2 coadministered with danicopan on Day 5.
  Treatment G1 (Period 2): 40 mg omeprazole administered once daily (QD) on Days 1-4.
  Treatment G2 (Period 2): 40 mg omeprazole administered QD with 200 mg danicopan administered orally TID on Days 5-8.
  There was a washout period of 2 days between the last dose of danicopan in Period 1 and the first dose of omeprazole in Period 2.
  Interventions: Drug: Danicopan; Drug: Calcium Carbonate; Drug: Aluminum/Magnesium Hydroxide/Simethicone; Drug: Omeprazole

INTERVENTIONS:
Drug: Danicopan — Oral tablet.
  Other Names: ALXN2040; ACH-0144471 (formerly); ACH-4471; ACH4471; 4471
Drug: Cyclosporine — Oral capsule.
  Other Names: Neoral
  Arms: Part 1: Danicopan plus Cyclosporine
Drug: Tacrolimus — Oral capsule.
  Other Names: Prograf
  Arms: Part 2: Danicopan plus Tacrolimus
Drug: Calcium Carbonate — Chewable tablet.
  Other Names: Antacid
  Arms: Part 3: Danicopan plus Antacids and Omeprazole
Drug: Aluminum/Magnesium Hydroxide/Simethicone — Chewable tablet.
  Other Names: Antacid; Gelusil
  Arms: Part 3: Danicopan plus Antacids and Omeprazole
Drug: Omeprazole — Oral, delayed-release capsule.
  Other Names: Prilosec
  Arms: Part 3: Danicopan plus Antacids and Omeprazole

SUMMARY:
This was a 3-part study with each part being an open-label, fixed-sequence, 2-period study in healthy adult participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index in the range of 18.0 to 32.0 kilograms (kg)/meter squared, inclusive, with a minimum body weight of 50.0 kg at Screening.
* Female participants must have been of non-childbearing potential and not needing to employ a method of contraception.
* Non-sterile male participants must have agreed to abstinence or used a highly effective method of contraception.
* No clinically significant history or presence of electrocardiogram findings at Screening and Day -1 of Period 1.

Key Exclusion Criteria:

* Evidence of any clinically significant deviation from normal in clinical laboratory evaluations.
* History of any medical or psychiatric condition or disease that might have limited the participant's ability to complete or participate in this clinical study, confound the results of the study, or pose an additional risk to the participant by their participation in the study.
* History or presence of drug or alcohol abuse within 2 years prior to first dosing; current tobacco/nicotine users and smokers; positive drugs-of-abuse and/or alcohol screen at Screening or Day -1 of Period 1.
* Any previous procedure that could have altered absorption or excretion of orally administered drugs.
* A history of significant multiple and/or severe allergies or had had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs.
* Body temperature ≥ 38°Celsius at Screening, on Day -1, or Day 1 prior to first dosing; history of febrile illness, or other evidence of infection, within 14 days prior to first dosing.
* Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 5 half-lives (if known) or 30 days before first dosing, whichever was longer.
* Donation of whole blood from 3 months prior to first dosing, or of plasma from 30 days before first dosing; receipt of blood products within 6 months prior to first dosing.
* Part 3 Only: Genotyped as poor metabolizer of cytochrome P450 2C19.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2018-10-17 (Actual)

PRIMARY OUTCOMES:
Part 1: Cyclosporine Maximum Observed Concentration (Cmax) Following Single-dose Cyclosporine Alone Versus In The Presence Of Steady-state Danicopan | Up to 72 hours postdose
Part 1: Cyclosporine Time To Reach The Maximum Observed Concentration (Tmax) Following Single-dose Cyclosporine Alone Versus In The Presence Of Steady-state Danicopan | Up to 72 hours postdose
Part 1: Cyclosporine Area Under The Concentration-time Curve From Time 0 Extrapolated To Infinity (AUC0-inf) Following Single-dose Cyclosporine Alone Versus In The Presence Of Steady-state Danicopan | Up to 72 hours postdose
Part 2: Tacrolimus Cmax Following Single-dose Tacrolimus Alone Versus In The Presence Of Steady-state Danicopan | Up to 144 hours postdose
Part 2: Tacrolimus Tmax Following Single-dose Tacrolimus Alone Versus In The Presence Of Steady-state Danicopan | Up to 144 hours postdose
Part 2: Tacrolimus AUC0-inf Following Single-dose Tacrolimus Alone Versus In The Presence Of Steady-state Danicopan | Up to 144 hours postdose
Part 3: Steady-state Omeprazole Cmax Following Multiple-dose Omeprazole Alone Versus In The Presence Of Steady-state Danicopan | Up to 24 hours postdose
Part 3: Steady-state Omeprazole Tmax Following Multiple-dose Omeprazole Alone Versus In The Presence Of Steady-state Danicopan | Up to 24 hours postdose
Part 3: Steady-state Omeprazole Area Under The Concentration-time Curve From Time 0 To The 24-hour Time Point (AUC0-24) Following Multiple-dose Omeprazole Alone Versus In The Presence Of Steady-state Danicopan | Up to 24 hours postdose
Part 3: Steady-state Danicopan Cmax Alone Versus In The Presence Of Multiple-dose Omeprazole | Up to 8 hours postdose
Part 3: Steady-state Danicopan Tmax Alone Versus In The Presence Of Multiple-dose Omeprazole | Up to 8 hours postdose
Part 3: Steady-state Danicopan Area Under The Concentration-time Curve From Time 0 To The 8-hour Time Point (AUC0-8) Alone Versus In The Presence Of Multiple-dose Omeprazole | Up to 8 hours postdose
Part 3: Steady-state Danicopan Cmax Alone Versus In The Presence Of Single-dose Calcium Carbonate Or Aluminum/Magnesium Hydroxide/Simethicone | Up to 8 hours postdose
Part 3: Steady-state Danicopan Tmax Alone Versus In The Presence Of Single-dose Calcium Carbonate Or Aluminum/Magnesium Hydroxide/Simethicone | Up to 8 hours postdose
Part 3: Steady-state Danicopan AUC0-8 Alone Versus In The Presence Of Single-dose Calcium Carbonate Or Aluminum/Magnesium Hydroxide/Simethicone | Up to 8 hours postdose

SECONDARY OUTCOMES:
Number Of Participants Experiencing Treatment-emergent Adverse Events | Day 1 through up to Day 31

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes